CLINICAL TRIAL: NCT03724851
Title: A Phase 1b/2a, Open-label, Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of Vactosertib in Combination with Pembrolizumab in Patients with Metastatic or Locally Advanced Colorectal or Gastric Cancer/ Gastroesophageal Junction Adenocarcinoma
Brief Title: Vactosertib in Combination with Pembrolizumab in Metastatic Colorectal or Gastric Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MedPacto, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP-VAC-204; Mk3475 Keynote 900 (Other: MSD)
Record Dates: First submitted 2018-10-10; First posted 2018-10-30 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Colorectal Cancer; Gastric Cancer; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms | interventions — vactosertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose Expansion (300mg BID) (Experimental): TEW-7197 300mg BID, 5D/W + Pembrolizumab 200mg Q3W (n= 30)
  Interventions: Drug: TEW-7197
- Dose Expansion (200mg BID) (Experimental): TEW-7197 200mg BID, 5D/W + Pembrolizumab 200mg Q3W (n= 30)
  Interventions: Drug: TEW-7197
- Dose Expansion (200mg QD) (Experimental): TEW-7197 200mg QD, 5D/W + Pembrolizumab 200mg Q3W (n= 30)
  Interventions: Drug: TEW-7197

INTERVENTIONS:
Drug: TEW-7197 — Vactosertib will be administered orally without regard to meals for 5 days per week (5D/W) at the same time in the morning (QD), at the same time in the morning and evening (BID) approximately 12 hours apart.
  Pembrolizumab will be administered as a dose of 200 mg using a 30-minute IV infusion. Sites should make every effort to target infusion timing to be as close to 30 minutes as possible.
  Other Names: vactosertib

SUMMARY:
This is an open-label, multicenter study to assess the safety, tolerability, pharmacokinetics, and antitumor activity of vactosertib in combination with pembrolizumab in patients with metastatic or locally advanced colorectal or gastric/gastroesophageal junction adenocarcinoma

DETAILED DESCRIPTION:
This is phase 1b/2a, open label, multi-center study to assess safety, tolerability, pharmacokinetics and anti-tumor activity of vactosertib in combination with pembrolizumab in patients with mCRC including CMS4 or diffuse GC/GEJC with two phases (Dose Finding Phase and Dose Expansion Phase). At screening, CMS4 will be classified by an experienced pathologist in the central lab that will examine the histology of primary surgical tissues. Approximately, 67 total patients are expected to be enrolled in this study. The first phase of the study, the Dose Finding Phase, will determine the MTD of the combination regimen. The second phase, the Dose Expansion Phase, will further evaluate the combination regimen to confirm RP2D.

ELIGIBILITY:
[Inclusion Criteria]

General Inclusion Criteria

1. Male and female Age ≥19 years at the time of screening
2. Patients must be able to swallow tablets and absorb vactosertib.

[Diagnosis/Condition for Entry into the Trial]

1. World Health Organization (WHO) / Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1 at enrollment
2. Must have a life expectancy of at least 12 weeks
3. Patients with histologically or cytologically confirmed advanced or metastatic non microsatellite instability high (MSI-H)/mismatch repair deficiency (dMMR) colorectal cancer who have disease progression after treatment with all available therapies including fluoropyrimidine and oxaliplatin or irinotecan for metastatic disease that are known to confer clinical benefit, or are intolerant to treatment, or refuse standard treatment.
4. Patients with histologically- or cytologically- confirmed, advanced or metastatic diffuse-type adenocarcinoma of the stomach or gastroesophageal (GE) junction who have had disease progression after at least two previous courses of chemotherapy for metastatic disease, which should include fluoropyrimidine and platinum.
5. Confirmation of measurable disease based on RECIST 1.1 by investigators at Screening will be used to determine patient eligibility and imaging shows at least 1 lesion that is appropriate for selection as a target lesion per RECIST 1.1 is required prior to patient treatment. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions. Tumor assessment by computed tomography (CT) scan or magnetic resonance imaging (MRI) must be performed within 28 days prior to C1D1.
6. All patients enrolled must be ICI-naïve patients defined as no prior exposure to immune-mediated therapy including, but not limited to, other anti CTLA-4, anti-PD-1, anti-PD-L1, and anti-programmed cell death ligand 2 (anti-PD-L2) antibodies, excluding therapeutic anticancer vaccines.
7. All patients must be able to provide a newly acquired tumor biopsy during screening (preferred) or provide an available archived tumor sample. Tumor lesions used for newly acquired biopsies should not be target lesions, unless there are no other lesions suitable for biopsy, and in this instance only core needle (not excisional/incisional) biopsy is allowed.
8. Patients must provide consent for an additional biopsy on C2D3-6 or C2D10-13. Post-treatment biopsy must be obtained from the same organ site as pre-treatment biopsy, if feasible, to avoid introduction of heterogeneity related to the site of tumor or metastasis. If submitting unstained cut slides, freshly cut slides should be submitted to the testing laboratory within 20 days from when the slides are cut. See Study Manual for an explanation.
9. Have adequate organ function as defined in the following Table 3.

[Exclusion Criteria]

Pregnancy Exclusion:

1. A woman of childbearing potential (WOCBP) who has a positive urine pregnancy test within 7 days prior to treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment.

Prior/Concurrent Clinical Study Experience

1. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

Prior/Concomitant Therapy

1. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137) Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks [could consider shorter interval for kinase inhibitors or other short half-life drugs] prior to treatment.
2. Has received prior radiotherapy within 2 weeks of start of study treatment. Patients must have recovered from all radiation-related toxicities, not require corticosteroids, and not 49 have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-central nervous system (CNS) disease.
3. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
4. The prohibited medications when using vactosertib are following (Refer to Appendix E). A minimal washout period of 5 half-lives for the following drugs is recommended prior to the first dosing.

Medical conditions

1. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 14 days prior the first dose of study drug.
2. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.

   Note: Patients with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, [additional examples can be added if important to the study such as transitional cell carcinoma of urothelial cancer], or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
3. Has known CNS metastases and/or leptomeningeal involvement
4. Has severe hypersensitivity (≥Grade 3) to pembrolizumab or vactosertib and/or any of its excipients
5. Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
6. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
7. Has an active infection requiring systemic therapy.
8. Has a known history of human immunodeficiency virus (HIV) infection or HIV test (+) in screening test. No HIV testing is required unless mandated by local health authority.
9. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.
10. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association Class III/IV), uncontrolled hypertension (≥150/90mmHg), unstable angina pectoris or myocardial infarction (≤ 6 months prior to screening), uncontrolled cardiac arrhythmia, clinically significant cardiac valvulopathy requiting treatment, active interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
11. QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥450 ms in male and ≥470 ms in female calculated from 12-lead ECGs
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | approximately 2 years
  Incidence of nature of DLTs
Safety and Tolerability | approximately 2 years
  Incidence, nature and severity of adverse events (AEs) graded according to NCI CTCAE v5.0

SECONDARY OUTCOMES:
Efficacy 1 | approximately 2 years
  Objective response rate (ORR) as assessed using RECIST version 1.1 and iRECIST by investigators
Efficacy 2 | approximately 2 years
  Progression Free Survival (PFS)
Efficacy 3 | up to 3 years
  Overall Survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Minkyu Heo, Study Director — MedPacto, Inc.
Locations (5):
- South Korea (5):
  - National Cancer Center, Goyang
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Yeonsei University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No